CLINICAL TRIAL: NCT05836337
Title: A Tattoo or a Clip? A Single-center Prospective Quasi Double-blind Randomized Parallel Two-arm Clinical Trial Evaluating the Effectiveness of a Tattoo Compared to a Clip Applied to Axillary Lymph Nodes in Breast Cancer Patients Who Undergo Sentinel Lymph Node Biopsy- SLNBx
Brief Title: Clinical Trial Evaluating the Effectiveness of a Tattoo Compared to a Clip Applied to Axillary Lymph Nodes in Breast Cancer Patients Who Undergo SLNBx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hussein Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16 KHCC 84
Record Dates: First submitted 2023-04-16; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a single-center prospective, randomized and quasi double blinded pilot study. The study includes 2 parallel arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tattoo- Black Eye (Experimental): to mark the biopsied axillary lymph node by tattooing
  Interventions: Device: Tattoo- Black Eye
- clip- HydroMARK (Active Comparator): To mark the biopsied axillary lymph node by clip placement
  Interventions: Device: clip- HydroMARK

INTERVENTIONS:
Device: Tattoo- Black Eye — Device name: Black eye Manufacturer: The Standard Co., Ltd
  Arms: Tattoo- Black Eye
Device: clip- HydroMARK — Device name: HydroMARK Manufacturer: Biopsy Sciences, LLC
  Arms: clip- HydroMARK

SUMMARY:
This study is a single-center prospective, randomized and quasi double blinded pilot study. The study has 2 parallel arms, each arm involved around 54 patients. Targeted community is the newly diagnosed adults with non metastatic and non inflammatory breast cancer in King Hussein Cancer Center who require axillary biopsy as part of their staging work up. The study aims to improve the intra-operative identification of the preoperatively suspicious and biopsied lymph nodes and test the concordance between the pre-operative clinical suspicion and histopathological results of these node; by comparing between preoperative marking of biopsied axillary lymph nodes with two different modalities (clipping Vs tattooing) and testing its concordance with sentinel lymph node biopsy, both in upfront surgery and neoadjuvant chemotherapy settings and in a prospective, randomized and quasi double blinded design

DETAILED DESCRIPTION:
This study is a single-center prospective, randomized and quasi double blinded pilot study. The study will enclose 2 parallel arms, each arm will involve 54 patients (total 108 patients), comparing between preoperative marking of biopsied axillary lymph nodes with two different modalities (clipping Vs tattooing) and testing its concordance with sentinel lymph node biopsy, both in upfront surgery and neoadjuvant chemotherapy settings and in a prospective, randomized and quasi double blinded design.

Targeted community is the newly diagnosed adults (more than 18 years of age) with non metastatic and non inflammatory breast cancer in King Hussein Cancer Center who require axillary biopsy as part of their staging work up.

The standards of breast cancer care in KHCC state that all patients are required to do breast and axillary staging via clinical examination and imaging (mammogram and U/S), and require any patient with clinically suspicious axillary lymph node/nodes to undergo U/S guided axillary biopsy. Patients with negative axillary biopsy will require axillary sentinel lymph node biopsy and patients having positive axillary lymph node biopsy will require axillary clearance along with their standard breast cancer surgical treatment.

Once the need for axillary biopsy is defined, the patients offered to participate in the study in a proper environment and their consent was gained after their approval. Participants were given another appointment few days later to obtain the axillary biopsy (as per the routine in the KHCC Breast Imaging Unit) and to mark the biopsied axillary lymph node in the same session, and on that day consented participants were randomized to either axillary lymph node clip placement or tattooing after obtaining the intended axillary biopsy.

Depending on the results of the biopsy, the KHCC breast MDC decided on the surgical management including the axillary treatment, the latter will be either sentinel lymph node biopsy (SLNBx)or axillary lymph node dissection (ALND). SLNBx will be performed on all recruited patients and to be followed by the standard axillary treatment as approved by KHCC clinical practice guidelines (either SLNBx alone or SLNBx followed by ALND). The group of patients with preoperative diagnosis of positive axillary nodes with undergo SLNBx as an extra procedure to test the study hypothesis and to be followed by ALND as per the KHCC protocol. The presence of the marking material will be confirmed prior to sending the SLNBx to the pathology department (by visualization of the tattoo and by X-ray examination of SLNBx looking for the clip). Patients whom receive ALND will have the presence of marking material checked in their specimens as well. This trial will study the concordance of both marking modalities with SLNBx identification

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosed with breast cancer.
* Scheduled for primary breast surgery with Sentinel Lymph node biopsy (SLNBx) or Axillary Lymph node dissection (ALND).
* Scheduled to undergo pre-operative axillary lymph node biopsy.
* Willing to sign the Informed Consent

Exclusion Criteria:

* Previous axillary surgeries, SLNBx and/or AD.
* Diagnosed with inflammatory breast cancer.
* Diagnosed with distant metastases.
* Known to have any allergic reaction to any of the investigational products.
* Participating in other studies involving investigational drug(s) (Phases 1-4) within 3 months prior to this study start and/or during study participation.
* Pregnant females or those with a positive pregnancy test result at screening or baseline; breastfeeding females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-08-20 (Actual)

PRIMARY OUTCOMES:
comparing effectiveness of tattooing versus clipping in SLNBx identification in breast cancer patients in upfront surgery setting, by comparing no. of identified positive or negative intraoperative SLN that were marked with tattooing versus clipping | 3 years
  To compare the effectiveness of tattooing compared to clipping in SLNBx identification in breast cancer patients in the upfront surgery and neoadjuvant setting, by comparing the number of identified positive or negative intraoperative SLN that were marked with the tattooing technique with the clip technique

SECONDARY OUTCOMES:
convenience for radiologist to apply clip or tattoo from time and technical perspectives by comparing time spent in applying clip or tattoo and convenience of the application using a questionnaire completed by radiologists after each application | 3 years
  The convenience for the radiologist to apply the clip or tattoo from time and technical perspectives by comparing time spent in applying the clip and tattoo as well as convenience of the application using a questionnaire completed by radiologists after each application
convenience for surgeon to perform SLNBx after lymph node marking from time & technical perspectives by comparing time and ease to identify the marked lymph nodes during surgery using a questionnaire completed by surgeons after each surgery | 3 years
  The convenience for the surgeon to perform the SLNBx after the lymph node marking from time and technical perspectives by comparing the time and ease to identify the marked lymph nodes during the surgery using a questionnaire completed by surgeons after each surgery
The convenience for the surgeon to confirm clip or tattoo presence during the SLNBx from time and technical perspectives using a questionnaire completed by surgeons after each surgery | 3 years
  The convenience for the surgeon to confirm clip or tattoo presence during the SLNBx from time and technical perspectives using a questionnaire completed by surgeons after each surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mahmoud Al-Masri, MD, Principal Investigator — King Hussein Cancer Center
Locations (1):
- King Hussein Cancer Center, Amman, Al 'A̅şimah, Jordan

IPD SHARING:
Plan to Share IPD: No